CLINICAL TRIAL: NCT04772339
Title: The Investigation of the Effects of Foot Core Muscles Endurance and Fatigue Resistance of These Muscles on Postural Stability and Gait Stability in Different Conditions
Brief Title: Effects of Foot Core Muscles Endurance and Fatigue on Postural Stability and Gait Stability
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Hilal Keklicek, Dr., Trakya University
Other Study IDs: TÜTF-BAEK 2019/101
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Gait Stability, Postural Stability
Keywords: Foot Core Muscles; Balance; Fatigue; Gait
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adults: Healthy adults aged between 18-30
  Interventions: Other: Heel-Rise Test; Other: Paper Grip Test (PGT)

INTERVENTIONS:
Other: Heel-Rise Test — The Heel Rise test for endurance will be performed while the participant stands on a box with 10 ° inclination on one leg. Participants will be allowed to get support from the wall at the point at shoulder level with two fingertips in order to maintain balance. A metronome of 30 beats per minute will be used to maintain the heel-rise frequency every 2 seconds. The participant will be asked to rise as high as possible with each heel rise, then lower the heel to the starting position, and with the next warning, he/she will be asked again. The participant will be asked to adapt to the pace of the metronome as much as possible and to continue the test as much as possible. The test will be terminated when the participant stops, fails to maintain frequency, or performs a proper heel raise. The number of heel raises obtained at the end of the test will be used for data analysis.
Other: Paper Grip Test (PGT) — In the paper grip test, a paper is placed under the individual's thumb and the person is asked to squeeze this paper strongly between the big toe and the ground. The paper is pulled by the person performing the test and the individual is asked to hold the paper with his/her thumb as much as he/she can. When the person applies the maximum force, the height of the medial longitudinal arch is measured with a digital caliper in millimeters. The time that the individual can maintain the MLA height with this maximum force is recorded with a stopwatch.

SUMMARY:
While walking, fatigue, sensorimotor function and motor control can affect in many ways. This research focuses on the relationship between foot core muscles with balance and gait parameters. The main purpose of the project is to investigate the effect of the endurance and fatigue responses of the extrinsic and intrinsic foot core muscles and the isolated fatigue response of the tibialis posterior muscle on balance and gait parameters.

DETAILED DESCRIPTION:
The foot core system is responsible for the stability and dynamic and static function of the foot. Foot core muscles are part of the sub-systems that make up this system. Fatigue affects the basic characteristics of the sensorimotor system and impairs the accuracy of the voluntary movement. While walking, fatigue, sensorimotor function and motor control can affect in many ways. This research focuses on the relationship between foot core muscles with balance and gait parameters. The main purpose of the project is to investigate the effect of the endurance and fatigue responses of the extrinsic and intrinsic foot core muscles and the isolated fatigue response of the tibialis posterior muscle on balance and gait parameters.

The method of the project was established to investigate the effects of foot core muscles on balance and gait parameters. Demographic and basic physical characteristics of the participants (age, dominant hand, height, weight, education, marital status) will be taken and individuals with normal BMI will be included in the study. Each individual will walk on the treadmill for at least 512 steps at the rate he/she will have at his own pace. Then the individual will rest. Then the gait test on the 10% slope will be repeated and the individual will rest at the end of the test. The balance of individuals' will be evaluated with Y balance test after the resting process is ended. The Heel Rise test will be used to measure the endurance of the tibialis posterior muscle. The test will be repeated separately for both feet. Then the individual will be put on the gait and balance tests. The individual will be recalled the next day and the paper grip test will be performed to measure the total endurance of the foot core muscles. Then the individual will be put on the gait and balance tests.

With this research; the relationship between the endurance and fatigue responses of the foot core muscles, which have an important role in the protection and support of the foot arches and which perform this function with tonic contraction in daily life, will be determined. In this way, the results of the research will provide information to explain the gait cycle. We believe that with an original study we may support the development of rehabilitation processes for individuals who have gait problems or who are at risk of falling.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 18-30
* Being within the limits of body mass index (weight / height2: 18.5-24.9 kg / m2) accepted as normal BMI by the World Health Organization
* To have the ability to speak and understand Turkish
* Agree to participate in the study

Exclusion Criteria:

* To be screened with any medical pre-diagnosis (orthopedic, neurological, cardiovascular, psychiatric, etc.)
* Being monitored with any medical diagnosis (orthopedic, neurological, cardiovascular, psychiatric etc.)
* Taking medication during the research
* Having consumed alcohol in the past 48 hours
* Taking pain medication in the past 48 hours
* Having a history of surgery or acute trauma in the last 6 months
* Having a fall for any reason within the last 1 year

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults aged between 18-30 within the normal BMI range by standards of WHO.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-04-08 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Gait analysis | It will be recorded at baseline, after the heel-rise test and after the paper-grip test
  Gait will be evaluated by a sensor gait analysis system. Sensors of this system are attached to the shoes of the individual and do not touch the skin. Each individual will freely walk on the treadmill for a period of time to achieve at least 512 steps at his/her own pace. To find the preferred walking speed of the individual, we will use the Hinton et al. protocol (Hinton et al., 2018). After the speed is determined, the individual will be provided to practice walking at this speed for 4-5 minutes. Then the walk will continue until at least 512 steps required for gait analysis are collected. After reaching the sufficient number of steps, the individual will be asked to slow down and stop walking. Then the individual will be taken to rest. The rest period will be determined according to the preference of the individual. Then the gait test will be repeated on 10% inclined ground and at the end of the test, the individual will rest again.
Y Balance Test | It will be recorded 5 minues after the gait analysis at baseline, after heel-rise test and after paper-grip test
  In the test setup, 3 length gauges (tape measure) are fixed on the non-slip surface to make an angle of 120 degrees with each other. The participant will be asked to stand on one leg of his/her choice at the intersection of these 3 measuring tapes, and to reach out with his/her toe in 3 directions with the other foot: anterior, posteromedial, and posterolateral. In the meantime, attention will be paid to ensure that the participant does not lose his balance, the heel of the foot on which he is standing does not rise from the ground, and the toes of the extended foot are just slightly touching the ground. This application will be repeated 3 times for each direction, averaged and recorded in cm, and the total score will be determined by proportioning the individual's functional leg length (trochanter major and ground distance).

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Faculty of Health Sciences, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No